CLINICAL TRIAL: NCT05811702
Title: The Impact of High-Fat Ketogenic Diet and Low-Fat Diet in the Body Weight and Cardiovascular Risk Factors on Overweight and Obese Saudi Women: A Randomized Controlled Trial.
Brief Title: The Impact of High-Fat Ketogenic Diet and Low-Fat Diet in Women Body Weight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal University (Other)
Responsible Party: Principal Investigator, Randah Miqbil Alqurashi, Assistant professor, King Faisal University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KingFaisalU
Record Dates: First submitted 2023-03-07; First posted 2023-04-13 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Overweight and Obesity; Healthy
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fat Ketogenic Diet (HFKD) (Experimental): A randomized acute controlled trial of twenty-eight healthy overweight or obese women in Saudi Arabia, aged between 18 and 40 with a body mass index between 25 and 34.5 kg m2 and fat parentage above 30% . The participants have followed ether HFKD for 12 weeks. The weight will be measured weekly, body fat % and blood samples before and after 12 weeks of following HFKD.
  Interventions: Other: A randomized acute controlled trial of twenty-eight healthy overweight or obese women
- low-fat diet (LFD (Experimental): A randomised acute controlled trial of twenty-eight healthy overweight or obese women in Saudi Arabia, aged between 18 and 40 with a body mass index between 25 and 34.5 kg m2 and fat parentage above 30% . The participants have followed ether LFD for 12 weeks. The weight will be measured weekly, body fat % and blood samples before and after 12 weeks of following LFD.
  Interventions: Other: A randomized acute controlled trial of twenty-eight healthy overweight or obese women

INTERVENTIONS:
Other: A randomized acute controlled trial of twenty-eight healthy overweight or obese women — A randomized acute controlled trial of twenty-eight healthy overweight or obese women in Saudi Arabia, aged between 18 and 40 with a body mass index between 25 and 34.5 kg m2 and fat parentage above 30% . The participants have followed ether HFKD or LFD for 12 weeks. Our primary outcome of this study to investigated the effective diets HFKD and LFD on reduction of body weight, the percentage of body fat

SUMMARY:
The aim of this study is investigated the effect of high fat Ketogenic Diet (HFKD) in weight reduction compared to the low-fat diet (LFD) among Saudi overweight and obese women. A randomized acute controlled trial of twenty-eight healthy overweight or obese women in Saudi Arabia, aged between 18 and 40 with a body mass index between 25 and 34.5 kg m2 and fat parentage above 30% . The participants have followed ether HFKD or LFD for 12 weeks.

DETAILED DESCRIPTION:
Obesity is associated with an increased risk of high blood pressure and heart muscle damage, which leads to cases that increase the chances of developing cardiovascular diseases, and if weight gain is not controlled, these results lead to obesity is the main cause of cardiovascular disease and causes dyslipidemia, high blood pressure and diabetes. Recently, there have been followed systems and programs food some of which are beneficial for health and some of them are unhealthy systems. The diet is one of the most controversial issues. The aim of this study is investigated the effect of high fat Ketogenic Diet (HFKD) in weight reduction compared to the low-fat diet (LFD) among Saudi overweight and obese women. A randomized acute controlled trial of twenty-eight healthy overweight or obese women in Saudi Arabia, aged between 18 and 40 with a body mass index between 25 and 34.5 kg m2 and fat parentage above 30% . The participants have followed ether HFKD or LFD for 12 weeks. Our primary outcome of this study to investigated the effective diets HFKD and LFD on reduction of body weight, the percentage of body fat, The secondary outcomes have evaluated at the percentage of body fat, blood glucose, lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Overwight and obese wonen
* aged 18 and 40
* BMI 25 and 34.5 kg m2
* fat parentage above 30% .

Exclusion Criteria:

* Man
* women in normal weight or BMI less than 25 and 34.5 kg m2
* Breastfeeding and pregnant women

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — A randomized acute controlled trial of twenty-eight healthy overweight or obese women in Saudi Arabia, aged between 18 and 40 with a body mass index between 25 and 34.5 kg m2 and fat parentage above 30%
Enrollment: 28 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Body weight (kg) and BMI | 12 weeks
  primary outcome of this study to investigated the effective diets HFKD and LFD on reduction of body weight, the percentage of body fat,
percentage of body fat | 12 weeks
  Primary outcome of this study to investigated the effective diets HFKD and LFD on reduction of percentage of body fat,

SECONDARY OUTCOMES:
Total Cholesterol mg/dl | 12 weeks
  Secondary outcome of this study to investigated the effective diets HFKD and LFD on total Cholesterol mg/dl
Triglycerides) mg/dl ( | 12 weeks
  Secondary outcome of this study to investigated the effective diets HFKD and LFD on total Triglycerides) mg/dl (
HDL) mg/dl ( | 12 weeks
  HDL) mg/dl (
LDL) mg/dl ( | 12 weeks
  LDL) mg/dl (
Glucose (mg/dl) | 12 weeks
  Glucose (mg/dl)
Hb Aic (%) | 12 weeks
  Hb Aic (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Randah Alqurashi, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No